CLINICAL TRIAL: NCT02543398
Title: Evaluation of Healing at Molar Extraction Sites With and Without Ridge Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Osteogenics Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20130470H
Record Dates: First submitted 2015-08-20; First posted 2015-09-07 (Estimated); Results first posted 2017-11-01 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2017-05

CONDITIONS: Loss of Teeth Due to Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ridge preservation (Other): The molar extraction socket is grafted with FDA approved materials, which includes a bone graft material derived from human donors (enCore®, Osteogenics biomedical, Lubbock, TX) and a membrane (like a thin sheet of paper) covering the grafted extraction socket. The membrane used will need to be removed at a later point since it is non-resorbable (it will not "dissolve" by itself). This membrane is made of dense polytetrafluoroethylene (dPTFE) (Cytoplast™, Osteogenics biomedical, Lubbock, TX). The procedure is called "Ridge preservation"
  Interventions: Procedure: Ridge preservation
- No ridge preservation (Other): The molar extraction socket is left to heal by itself without any grafting material or membrane, i.e. "Spontaneous Healing" (No ridge preservation is performed)
  Interventions: Procedure: Ridge preservation

INTERVENTIONS:
Procedure: Ridge preservation — Ridge preservation is a procedure which consists in grafting the tooth extraction socket with a bone grafting material and cover the site with a membrane to protect the site.

SUMMARY:
Following tooth extraction ridge preservation procedure have been suggested to limit bone resorptive dimensional changes to facilitate prospective implant placement. While this is particularly true for anterior teeth, no evidence is available to establish clinical guidelines in posterior sites, i.e. following molar extraction.

This research project will answer the following question:

What are the dimensional changes of the hard and soft tissues encountered following molar extractions with and without ridge preservation?

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included in this study if they qualify the following inclusion criteria:

  * One molar tooth that has been identified by dental faculty as requiring a single tooth extraction
  * A dental implant is indicated and treatment planned to replace the missing molar tooth
  * Have adequate restorative space for a dental implant-retained restoration
  * Have at least 10mm of alveolar bone height, without impinging on the maxillary sinus or inferior alveolar canal.

Exclusion Criteria:

* Obvious exclusions are patients who do not meet all the inclusion criteria or who will not cooperate with the follow-up schedule.
* Patients will not be entered who are mentally incompetent, prisoners, or pregnant.
* Pregnant women or women intending to become pregnant during the study period. As standard practice prior to dental surgery, females of child-bearing age are asked verbally if there is any possibility that they are pregnant. If not, we proceed with surgery and no pregnancy test is done. If the woman states that there is a possibility that she is pregnant, we do a urine pregnancy test to rule pregnancy in or out. So use of the urine pregnancy test is only done if she says she may be pregnant. [If needed: An over-the-counter urine pregnancy test will be provided to female subjects in the graduate periodontics clinic of UTHSCSA. Patients will be allowed access to a private restroom and the results of the tests will be read by one of the named investigators. Only those with a negative pre-operative pregnancy test will be eligible for the study.] Female patients who have undergone a hysterectomy, tubal ligation or menopause will be excluded from pregnancy testing.
* Patients who become pregnant during the study will be withdrawn and standard care will be delivered.
* Clinical and/or radiographic determinations which will preclude inclusion in this study are:

  * Active localized or systemic infection other than periodontitis.
  * Untreated periodontal diseases
  * Inadequate bone dimensions or restorative space dimensions to place a dental implant
  * Presence of a disease entity, medical condition or therapeutic regimen which decreases probability of soft tissue and bony healing, e.g., poorly controlled diabetes, chemotherapeutic and immunosuppressive agents, or autoimmune diseases.
  * Positive medical history of endocarditis following oral or dental surgery.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-10; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

REFERENCES:
- [Derived] Walker CJ, Prihoda TJ, Mealey BL, Lasho DJ, Noujeim M, Huynh-Ba G. Evaluation of Healing at Molar Extraction Sites With and Without Ridge Preservation: A Randomized Controlled Clinical Trial. J Periodontol. 2017 Mar;88(3):241-249. doi: 10.1902/jop.2016.160445. Epub 2016 Oct 27. PMID 27788625

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Location: Graduate Periodontics clinic at the University of Texas Health Science Center at San Antonio (UTHSCSA), San Antonio, Texas Date: January 2014 to May 2015
Period: Overall Study
Arm/Group | Ridge Preservation | No Ridge Preservation
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ridge Preservation | No Ridge Preservation | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (11.5) | 53.3 (10.7) | 53.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 13 | 13 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Bone Changes
Description: The width and the height of the alveolar ridge will be measured (in mm) on the initial (i.e. following tooth extraction) Cone Beam CT and on the CBCT taken prior to implant placement (i.e. 3 months after tooth extraction)
Time Frame: 3 months after tooth extraction
Measure: Mean (Standard Error); unit: millimeter
Arm/Group | Ridge Preservation | No Ridge Preservation
Number analyzed (Participants) | 20 | 20
millimeter
  Bone height change | -1.12 (1.60) | -2.60 (2.06)
  Bone width change | -1.16 (1.97) | -.158 (2.23)

ADVERSE EVENTS:
Time Frame: Data were collected until study completion that is when the patient received their dental implant
Arm/Group | Ridge Preservation | No Ridge Preservation
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No